CLINICAL TRIAL: NCT03502018
Title: Evaluation of the Efficacy of Exparel Delivered Into the Hip Capsule During Hemiarthroplasty
Brief Title: Hip Fracture Exparel Administration Trial Capsule During Hemiarthroplasty
Acronym: HEAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Kevin Kang, Primary research investigator, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-10-01
Record Dates: First submitted 2018-03-27; First posted 2018-04-18 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Intracapsular Fracture of Femur; Femoral Neck Fractures; Hip Hemiarthroplasty
Keywords: Exparel; Bupivacaine; Intracapsular Fracture of the Femur; Femoral Neck Fracture; Hip Hemiarthroplasty
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: There will be a total of 50 patients enrolled in this randomized blinded prospective two arm study. The participants will be randomized into either the control or the EXPAREL treatment group, with 25 patients in each cohort.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, Investigator(s), outcome assessors will all be blinded throughout the duration of the trial. Care providers pre- and post- op will be blinded as well, the operative team will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline (Placebo Comparator): This arm will receive Saline along with Bupivacaine
  Interventions: Drug: Saline
- Bupivacaine liposome (Experimental): This arm will receive Exparel along with Bupivacaine
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Bupivacaine liposome — A long-acting liposomal bupivacaine
  Other Names: Exparel
  Arms: Bupivacaine liposome
Drug: Saline — Saline injection used as control
  Other Names: No other names
  Arms: Saline

SUMMARY:
This study will examine the efficacy of Liposomal Bupivacaine (Exparel) in hip fracture patients undergoing hip hemiarthroplasty for femoral neck fractures through a posterior approach. Post-operative measures will be assessing pain, overall opiate use, delirium, time-to-ambulation and discharge status.

DETAILED DESCRIPTION:
Exparel is a long-acting and sustained release formulation of the local anesthetic, bupivacaine HCl. Recent studies have supported its efficacy following total joint arthroplasty, but little is known about Exparel's effectiveness in hip fracture patients. This investigation will study the effects of Exparel on postoperative pain following hip fracture surgery. This is a single center, randomized prospective double blinded study of 50 patients with hip fractures that will have intracapsular hip hemiarthroplasties and are 65 years or older. Twenty-five patients will be treated with intraoperative injections of Exparel. Current standard of care does not include any injection of pain medication during hip hemiarthroplasty. There is no 'standard treatment', but to use multimodal IV and oral analgesia. The control group consisting of the remaining 25 patients will receive 'standard treatment' (which is is multimodal IV and oral analgesia). Therefore, saline is the appropriate placebo and control injection for this study. There are minimal to no risks associated with the injection of saline into the soft tissues about the hip and will take <2 minutes to complete. The surgeries will be performed by five surgeons who will use their standard treatment or in the interventional group participants will relieve 20 cc of Exparel diluted with 40 ml 0.25% bupivacaine into the surrounding hip capsule: external rotators, gluteus medius, gluteus minimus, gluteus maximus, tensor fascia lata, vastus lateralis, and subcutaneous tissues.

Both the patient and the researcher following the patient postoperatively will be blinded. While the treating surgeon will be able to notice the difference between the placebo and Exparel, the outcomes outlined below will be recorded by the blinded Orthopaedic Research Resident who has no clinical responsibilities during his/her year of research and does not participate in operative procedures

There are two overall aims of this investigation. The first aim is to identify whether Exparel has an impact on postoperative pain and function following open treatment of hip fractures. The hypothesis is that injecting Exparel into the hip capsule and surrounding tissues will decrease narcotic use, and in turn decrease the risk of associated side effects including medically induced delirium, constipation, and decreased alertness. The second aim of the study is focused on examining whether increased pain control leads to better postoperative outcomes? When pain is better controlled via non-narcotic measures, overall patient comfort will improve while sparing cognitive function, decreasing time to ambulation, and accelerating progress with physical therapy. Quicker recovery times will then produce shorter hospital stays, which would yield better overall patient satisfaction and overall improved outcomesPatients with intracapsular hip fractures will undergo hip hemiarthroplasty using a bipolar prosthesis placed via a posterior approach. Primary outcome measures include postoperative visual analogue scale (VAS from 0-10) pain scores at 12, 24, 36, 48 hours after surgery, time to ambulation with physical therapy, need for postoperative total morphine equivalent, and delirium scale measurements. Secondary outcomes measures will compare length of stay, discharge disposition (home or skilled nursing facility), 30-day readmission rates, and adverse events leading to ICU care or reoperation. All patients in both groups will have access to breakthrough pain medication which will either be Immediate acting Oxycodone for moderate to severe pain (pain scale of 4-10, Acetaminophen or Toradol for mild to moderate pain (pain scale of 2-4).

ELIGIBILITY:
Inclusion Criteria:

Men and women sixty-five years of age and older with isolated intracapsular hip fractures undergoing hemi arthroplasty through a posterior approach with the ability to consent to the study.

Exclusion Criteria:

Under sixty-five years of age, extracapsular hip fracture, suffer from any form of cognitive compromise that leaves them unable to consent, or if they are treated with any surgical modality other than hip hemiarthroplasty.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Komlos, MD, PhD, Principal Investigator — Maimonides Medical Center; Kevin Kang, MD, Study Director — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline | Bupivacaine Liposome
Started | 25 | 25
Completed | 24 | 25
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | Bupivacaine Liposome | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 24 | 25 | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 4 | 7 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 16 | 23 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 49

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain
Description: Primary outcome measure will be postoperative visual analogue scale (VAS from 0-10) pain scores. 0 = no pain, 10 = most pain
Time Frame: 4hrs after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
score on a scale | 3.29 (2.66) | 2.64 (2.27)

2. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 8hrs after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
score on a scale | 3.04 (1.64) | 2.12 (1.79)

3. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 12hrs after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
score on a scale | 2.42 (2.19) | 2.08 (2.72)

4. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 24hrs after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
score on a scale | 2.58 (2.86) | 2.00 (2.48)

5. Primary Outcome: Post-operative Pain
Description: as for outcome 1
Time Frame: 48hrs after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
score on a scale | 2.71 (3.10) | 2.04 (2.69)

6. Secondary Outcome: Time to Ambulation
Description: Measure of time to ambulation with physical therapy
Time Frame: 24 and 48 hours after surgery
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
Days | 1.44 (0.82) | 1.12 (0.53)

7. Secondary Outcome: Postoperative Total Morphine Equivalent
Description: Total dose in milligrams of opiates measured in total morphine equivalents. This was measured by calculating the sum of total morphine equivalents administered within 48 hours postoperatively. Assessed at 12, 24, 36, 48 hours after surgery, total postoperative total morphine equivalents at 48 hours after surgery reported
Time Frame: 48 hours after surgery
Measure: Mean (Standard Deviation); unit: Morphine Equivalent
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
Morphine Equivalent | 9.98 (10.638927) | 12.09 (9.65)

8. Secondary Outcome: Delirium Scale Measurements
Description: Assessment of post-operative delirium based on Short Confusion Assessment Method
Time Frame: 24 and 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
Participants
  At 24 Hours | 0 | 1
  At 48 Hours | 0 | 0
  No Delirium | 24 | 24

9. Secondary Outcome: Length of Stay
Description: Total days until discharge from hospital
Time Frame: 7 days from day of admission
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Saline | Bupivacaine Liposome
Number analyzed (Participants) | 24 | 25
Days | 3.88 (2.13) | 3.92 (1.44)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of surgery until the 30 days postoperatively from 2018 to 2023
Arm/Group | Saline | Bupivacaine Liposome
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03502018/Prot_SAP_000.pdf